CLINICAL TRIAL: NCT02771613
Title: Impact on Adverse Events (AE) Occurrence of Two Types of Experience Feedback on AE Analysed During Local Morbidity Mortality Reviews (MMR), (by Multi Professional Simulation Education Versus Simple Diffusion of MMR Decisions)
Brief Title: Impact on the Adverse Event (AE) Incidence of Two Types of Experience Feedback on AE Analyzed During Local Morbidity Mortality Reviews
Acronym: RMM Simulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0093
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Hospital Adverse Event
Keywords: Morbidity Mortality Review; medical simulation; in situ simulation; multi professional simulation; hospital adverse event

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Active experience feedback: Multi professional, in situ simulation , with scenarios based on the adverse events analyzed in MMR : After analysis of adverse effects in Morbidity Mortality reviews, we will create scenarios adapted to these events. Education of the randomized department's arm's staff will be performed by multi professional in situ simulation with these scenarios
  Interventions: Other: Multi professional in situ simulation
- Passive experience feedback: Large diffusion of information about discussions and decisions of Morbidity Mortality Reviews : after the analysis of adverse effects in Morbidity Mortality reviews, a large scale dissemination activity of information about discussions and decisions towards the staff of the randomized departments' arms will be carried out.
  Interventions: Other: Large diffusion of information
- No experience feedback: MMR will be performed as usual, without any feedback to the medical staff

INTERVENTIONS:
Other: Multi professional in situ simulation — After the analysis of adverse effects in Morbidity Mortality reviews, we will create scenarios adapted to these events. Education of the randomized department's arm's staff will be performed by multi professional in situ simulation with these scenarios
  Groups: Active experience feedback
Other: Large diffusion of information — After the analysis of adverse effects in Morbidity Mortality reviews a large scale dissemination activity of information about discussions and decisions towards the staff of the randomized departments' arms will be carried out
  Groups: Passive experience feedback

SUMMARY:
After implementing a French version of a trigger tool validated for computerized detection of adverse events in patient's medical record, the study will be performed in three parallel randomized arms of three identical departments (each steaming from 6 types of medical, surgical or obstetrical departments with a total of 18 departments involved). This three arms will be: no intervention, education of department's staff by multi professional in situ simulation (adapted to the discovered adverse events), or simple but large diffusion of results and decisions of Morbidity Mortality Reviews.

The interventions will be performed during a two-years period.

ELIGIBILITY:
Inclusion Criteria:

* patients aged > 18 years old
* patients hospitalized in the involved departments during the two-years intervention's period

Exclusion Criteria:

* patient aged < 18 years old
* no other exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: any stage of patients in the involved departments during the two-years intervention's period
Sampling Method: Non-Probability Sample
Enrollment: 144000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Occurence of adverse events related to medical care | During patient hospitalization, up to 2 years
  Occurrence of any adverse effects detected by the trigger tool. Trigger tool is used to detect more patient's adverse events that voluntary medical report

SECONDARY OUTCOMES:
Severity of adverse events related to medical care | During patient hospitalization, up to 2 years
  Severity of any patient's adverse effect detected by trigger tool. Severity of adverse events is measured by a severity score scale.
Contributive factors identification | During patient hospitalization, up to 2 years
  Contributive factors of adverse events using the "ALARM Method". The Alarm Method allows to determine the contributive factors which together create the adverse patients events.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard BUI-XUAN, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Direction DOQRU, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michel N, Bui-Xuan B, Bapteste L, Rimmele T, Lilot M, Chollet F, Favre H, Duclos A, Michel P. Implementation of an in situ simulation-based training adapted from Morbidity and Mortality conference cases: effect on the occurrence of adverse events-study protocol of a cluster randomised controlled trial. Trials. 2022 Feb 2;23(1):106. doi: 10.1186/s13063-022-06040-2. PMID 35109900